CLINICAL TRIAL: NCT03112759
Title: Assessing the Utility of Cognitive Behavioral Therapy for Pain Control in Patients With Chronic Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Gary C. Vitale, MD, General Surgeon, Professor of medicine, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17.0352
Record Dates: First submitted 2017-04-07; First posted 2017-04-13 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into one of two arms: treatment with cognitive behavioral therapy and narcotics as needed or treatment with conventional narcotic analgesics alone. Patients undergoing CBT intervention will participate in eight weekly therapy sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy (Experimental): Patients randomly selected for CBT will attend 8 weekly one-on-one therapy sessions. Patients will be prescribed conventional narcotic therapy as needed.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- No Cognitive Behavioral Therapy (No Intervention): Patients randomly selected for no CBT will be treated with conventional narcotic therapy alone.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Cognitive behavioral therapy (CBT) uses pain coping skills as a method of managing symptoms associated with chronic pain.Cognitive behavioral therapy teaches patients to identify and modify negative thoughts and behaviors that increase pain intensity, distress, and pain-related disability
  Arms: Cognitive Behavioral Therapy

SUMMARY:
This study will assess cognitive behavioral therapy as an adjunct to conventional symptom control for patients with chronic pancreatitis.

DETAILED DESCRIPTION:
All patients with chronic pancreatitis will be considered for participation in this study. Patients selected for participation will be evaluated 4 weeks prior to the first one-on-one therapy session. A baseline pain score will be assessed using the visual analog pain scale. Narcotic dosage and frequency as well as anti-emetic usage will be evaluated at this time. A pre-treatment quality of life score will be recorded using the SF-12® Patient Questionnaire. Patients will also be queried about the presence of nausea and reflux.

After the pre-intervention evaluations are complete, patients will be randomized into one of two arms: treatment with cognitive behavioral therapy and narcotics as needed or treatment with conventional narcotic analgesics alone. Patients undergoing CBT intervention will participate in eight weekly therapy sessions. Follow-up assessments will be conducted six months and nine months after the last therapy session is completed. The patients will be evaluated based on pain score, narcotic dosage and frequency, anti-emetic usage, quality of life assessment, and pain related hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be18 years of age
2. Diagnosed with chronic pancreatitis
3. Willing and able to comply with the protocol requirements
4. Able to comprehend and have signed the Informed Consent Form (ICF) to participate in the study

Exclusion Criteria:

1. Participating in another clinical trial for the treatment of chronic pancreatitis at the time of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-09-09 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

PRIMARY OUTCOMES:
Presence and severity of abdominal pain | 1 year
  A visual analog scale will be used to measure patients pain pre- and post- intervention

SECONDARY OUTCOMES:
Quality of Life | 1 year
  quality of life with be measured using the SF-12® Patient Questionnaire
Narcotic Usage | 1 year
  Narcotic usage will be monitored at each follow-up.
Presence and Severity of Nausea and Reflux | 1 year
  patients will be queried about the presence and severity of nausea and reflux at each follow-up appointment
Hospitalizations | 1 year
  Pre- and post- intervention hospitalizations will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yadav D, Lowenfels AB. The epidemiology of pancreatitis and pancreatic cancer. Gastroenterology. 2013 Jun;144(6):1252-61. doi: 10.1053/j.gastro.2013.01.068. PMID 23622135
- [Background] Gachago C, Draganov PV. Pain management in chronic pancreatitis. World J Gastroenterol. 2008 May 28;14(20):3137-48. doi: 10.3748/wjg.14.3137. PMID 18506917
- [Background] Heapy AA, Stroud MW, Higgins DM, Sellinger JJ. Tailoring cognitive-behavioral therapy for chronic pain: a case example. J Clin Psychol. 2006 Nov;62(11):1345-54. doi: 10.1002/jclp.20314. PMID 16937347
- [Background] Erdek MA, Pronovost PJ. Improving assessment and treatment of pain in the critically ill. Int J Qual Health Care. 2004 Feb;16(1):59-64. doi: 10.1093/intqhc/mzh010. PMID 15020561